CLINICAL TRIAL: NCT04440215
Title: Optimizing Patient Adherence to Stroke Rehabilitation Treatment: a Telerehabilitation Trial
Brief Title: Optimizing Patient Adherence to Stroke Rehabilitation Treatment
Acronym: Telestroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Collaborators: Université de Montréal (Other); Laval University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Isabelle Gaboury, Professor, Université de Sherbrooke
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: MP-04-2020-519
Record Dates: First submitted 2020-06-12; First posted 2020-06-19 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Stroke Rehabilitation; Telerehabilitation; Decision Making, Shared
Keywords: Rehabilitation; Stroke; Adherence; Home; Telerehabilitation; Interprofessional shared decision making
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: An interrupted time series design. It consists of observing the same dependent variable over time, with a break in the series of observations corresponding to the introduction of an intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Usual rehabilitation care (no telerehabilitation, interdisciplinary meetings not systematically organized and/or not involving a complete team of professionals)
  Interventions: Other: Usual care
- Telerehabilitation (Experimental): A mix of home or rehabilitation center visits, telerehabilitation and interprofessional shared decision making process.
  Interventions: Other: Telerehabilitation and team meetings and team care plans

INTERVENTIONS:
Other: Telerehabilitation and team meetings and team care plans — A mix of home or rehabilitation center visits and telerehabilitation will be planned by the rehabilitation team for a maximum of 16 weeks. Moreover, for each participant enrolled, a multidisciplinary meeting will be organised. The patient/family will participate in the meeting and the decision making process using the telerehabilitation platform. The team will generate an interprofessional individualized treatment plan, aiming for an interprofessional shared decision making process.
  Arms: Telerehabilitation
Other: Usual care — Rehabilitation teams will be instructed to provide care as they have been doing previously. Currently, this translates into no telerehabilitation, and interdisciplinary meetings not systematically organized and/or not involving a complete team of professionals.
  Arms: Control

SUMMARY:
Stroke impacts nearly 400,000 Canadians annually. Three quarters of stroke survivors will live with minor to severe impairments or disabilities; which require rehabilitation care. Strong evidence supports beginning rehabilitation as soon as the patient's medical status has stabilized and continuing following discharge from acute care. Access to optimal services is hampered, however, by travel distances to access rehabilitation, the lack of opportunities for structured and formal interprofessional communication among service providers, and failures to engage the patient and family members in a structured decision making process. Moreover, adherence to rehabilitation treatments has been shown to be suboptimal. Many patients refuse their outpatient rehabilitation treatments outright or decrease the duration and/or frequency of their treatments over time.

The aim of this proposed mixed methods pragmatic clinical trial is to evaluate an intervention that provides patients who have experienced stroke the opportunity to return home safely after their acute hospital stay, to encourage patient (and family) engagement in their rehabilitation care, and to overcome challenges of access to patient-centered interprofessional rehabilitation care.

The proposed intervention will entail 220 patients (and family) to receive rehabilitation care through remote, live treatment sessions with an interdisciplinary group of clinicians (called telerehabilitation) versus standard of care (n = 110 patients). Five rehabilitation teams will be trained to develop rehabilitation treatment plans that engage the patient and family, while taking advantage of a telerehabilitation platform to engage the patient/family. Grounded in findings gathered through a Canadian Institute of Health Research (CIHR) funded pilot study, the primary study objective is to evaluate process, clinical outcomes and costs of telerehabilitation in comparison with usual care. Through qualitative interviews with patients and family as well as clinicians, a second objective of this pragmatic, controlled trial is to explore and describe contextual factors (both personal and environmental) that will help the delivery of care, and improve patient's outcomes while fully using technology to deliver stroke rehabilitation care.

This study represents a unique, highly relevant opportunity to minimize both knowledge and practice gaps, while producing robust, indepth data on the factors related to the effectiveness of telerehabilitation.

DETAILED DESCRIPTION:
Stroke impacts nearly 400,000 Canadians annually. Three quarters of stroke survivors will live with minor to severe impairments or disabilities; which require rehabilitation care representing >$3.6 billion in Canadian healthcare expenditure every year. Strong evidence supports beginning rehabilitation as soon as the patient's medical status has stabilized and continuing following discharge from acute care, ideally in the patient's community. Access to optimal services is hampered, however, by travel distances to access rehabilitation, the lack of opportunities for structured and formal interprofessional communication among service providers, and failures to engage the patient and family members in a structured decision making process. Even when travel is not a barrier, adherence to rehabilitation treatments has been shown to be suboptimal. Many patients refuse their outpatient rehabilitation treatments outright or decrease the duration and/or frequency of their treatments over time.

The aim of this proposed mixed methods pragmatic clinical trial is to evaluate an intervention that provides patients who have experienced stroke the opportunity to return home safely after their acute hospital stay, to encourage patient (and family) engagement in their rehabilitation care, and to overcome challenges of access to patient-centered interprofessional rehabilitation care.

The proposed intervention will entail 220 patients (and family) to receive rehabilitation care through remote, live treatment sessions with an interdisciplinary group of clinicians (called telerehabilitation) versus standard of care (n = 110 patients). Five rehabilitation teams will be trained to develop rehabilitation treatment plans that engage the patient and family, while taking advantage of a telerehabilitation platform to engage the patient/family. Grounded in findings gathered through a CIHR funded pilot study, the primary study objective is to evaluate process, clinical outcomes and costs of telerehabilitation in comparison with usual care. Through qualitative interviews with patients and family as well as clinicians, a second objective of this pragmatic, controlled trial is to explore and describe contextual factors (both personal and environmental) that will help the delivery of care, and improve patient's outcomes while fully using technology to deliver stroke rehabilitation care.

This application has been developed by an interdisciplinary team of researchers, local healthcare providers from each region involved, two patient partners who have experienced stroke, provincial network stakeholders, and decision makers, all engaged in the successful implementation of stroke guidelines and jurisdictional strategic plans. A panel of Canadian health system knowledge users rounds out the team, to enhance the proposed intervention, to communicate the relevance and anticipated use of the findings within their province, and to foster adaptation of improved stroke care elsewhere. Finally, the study has been endorsed by several knowledge users from the Quebec Ministry of Health as well as the Quebec Heart and Stroke Foundation. Considering contrasts between rehabilitation practices and the Canadian Stroke recommendations and the lack of relevant, robust data, this study represents a unique, highly relevant opportunity to minimize both knowledge and practice gaps, while producing robust, indepth data on the factors related to the effectiveness of telerehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Have had stroke event (haemorrhagic or ischemic)
* Are considered to be safe for home discharge by the acute/ in-patient care team (i.e. mild to moderate Functional Independence Measure score)
* Have a relative or informal caregiver who is present in the home should physical rehabilitation treatments are required;
* Can speak French or English.

Exclusion Criteria:

* Having severe cognitive decline prior to the stroke event

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient adherence to stroke rehabilitation plan (Patient journal) | Through intervention completion (up to 12 weeks)
  Time spent (in minutes) doing any stroke rehabilitation exercises (online + offline). This includes (but is not limited to) physical, writing and speech therapy, and mental health-related exercises recommended by the rehabilitation professional.
Change in patient adherence to stroke rehabilitation plan | Change from baseline and 4-, 6-, 12-week post-recruitment
  StREAM questionnaire which is a 12-item questionnaire coted on a 4-point Likert scale which measure patients' adherence to a rehabilitation program.
Patient adherence to stroke rehabilitation plan (Professional perception) | Through intervention completion (up to 12 weeks)
  Health care professional perception of the participants' adherence to the rehabilitation program, evaluated on a 10-point scale.

SECONDARY OUTCOMES:
Sociodemographic questionnaire | At recruitment (baseline)
  Home questionnaire including information about sex, age, clinical information about stroke
Change in functional recovery and independence | Change from baseline and 12-week post-recruitment
  The modified 5-level Functional Independence Measure (FIM; 18 items) will be used. This measurement tool explores an individual's physical, psychological and social function. The tool is used to assess a patient's level of disability as well as change in patient status in response to rehabilitation or medical intervention. A lower score reflects greater disability.
Change in reintegration into normal social activities | Change from baseline and 12-week post-recruitment
  The Reintegration to Normal Living Index (RNLI; 11 items) will be used to assess the degree to which the participants perceived their normal social activities have been impacted by the stroke event. A higher score indicates more difficulty to reintegrate normal living.
Change in depression state | Change from baseline and 12-week post-recruitment
  The Beck Depression Inventory (Beck; 21 items) will be used to measure the severity of depression. The inventory is composed of items relating to depressive symptoms. A higher score indicates higher depression state.
Use of healthcare services | within 12 week and 6 month post recruitment
  This outcome, defined as expenses related to services and long-term complications, including hospitalization and physician visits is measured with 3 different tools: 1) Section A - Use of healthcare services (16 items) of the questionnaire developed by the Institut National de Santé Publique du Québec (INSPQ), 2) information collected daily by the participant in a calendar and 3) Health administrative provincial data on use of public health services received.
Adverse events | Through intervention completion (up to 12 weeks)
  Presence of adverse events related to rehabilitation (pain, dizziness, fatigue, number of falls)
Perception of interprofessional care shared decision making (Patient POV) | 12 weeks after recruitment
  The Collaboration and Satisfaction About Care Decision tool (9 items) will be used. This questionnaire will be completed by the health care professionals involved in the study.
Perception of interprofessional care shared decision making (Clinical team POV) | Through study completion (up to 5 years)
  The Assessment of Interprofessional Team Collaboration Scale, short version (AITCS; 23 items) will be used. This questionnaire will be completed by the health care professionals involved in the study.
Statistics related to the telerehabilitation platform use | Through intervention period (up to 3 years)
  Home questionnaire on telerehabilitation platform utilisation (who, when, duration).
Presence of intervention plan in the patient file | 12 weeks after recruitment
  A "Yes" or "No" answer to the presence of an intervention plan in the patient file
Specific shared decision making (SDM) behaviours during decision-making (Questionnaire) | At the start of the rehabilitation period
  A composite questionnaire (SURE, 4 questions; Assumed role for decision-making, 1 question; CollaboRATE, 3 questions; Quality in decision-making, 6 questions) will be used to assess the extent to which practitioners involve patients in decision making processes. Patients will be given this questionnaire following the meeting to establish their rehabilitation plan.
Specific shared decision making (SDM) behaviours during decision-making (Interviews) | At the start of the rehabilitation period
  A randomized sample of 60 patients will be selected (50% control, 50% intervention). The meetings to establish their treatment plan will be recorded and analyzed using qualitative methods, in order to document the dynamics of the decision-making process. This qualitative section of the study will help enrich and contextualize the quantitative data collected for the other outcomes.

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Centre de réadaptation en déficience physique - Installation Châteauguay, Châteauguay, Quebec
  - Centre de réadaptation en déficience physique - Installation Granby, Granby, Quebec
  - Centre de réadaptation en déficiences physique - Installation Saint-Hubert, Longueuil, Quebec
  - Centre de réadaptation en déficience physique - Installation Longueuil, Longueuil, Quebec
  - Centre de réadaptation en déficience physique - Installation Saint-Hyacinthe, Saint-Hyacinthe, Quebec
  - Centre de réadaptation en déficience physique - Installation Vaudreuil-Dorion, Vaudreuil-Dorion, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaboury I, Tousignant M, Corriveau H, Menear M, Le Dorze G, Rochefort C, Vachon B, Rochette A, Gosselin S, Michaud F, Bollen J, Dean S. Effects of Telerehabilitation on Patient Adherence to a Rehabilitation Plan: Protocol for a Mixed Methods Trial. JMIR Res Protoc. 2021 Oct 28;10(10):e32134. doi: 10.2196/32134. PMID 34709196